CLINICAL TRIAL: NCT02275806
Title: A Phase II Study of Definitive Concurrent Radiation Therapy With Cisplatin and Irinotecan Chemotherapy in Locally Advanced In-operable Non-Small Cell Lung Cancer
Brief Title: Cisplatin/Irinotecan With Concurrent Radiation for Inoperable NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI decided to terminate study
Sponsor: Leo W. Jenkins Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LJCC 2014-01
Record Dates: First submitted 2014-10-22; First posted 2014-10-27 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2018-10

CONDITIONS: Lung Neoplasms, Non-Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Irinotecan; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All enrolled patients (Other): Induction Chemotherapy Cycle 1 - Irinotecan 65 mg/m2 and Cisplatin 30 mg/m2 on days 1 and 8
  Concurrent Chemotherapy Cycles 2-4 - Irinotecan 65 mg/m2 and Cisplatin 30 mg/m2 on days 22 and 29, days 43 and 50, and days 64 and 71 along with radiation therapy of 60-70 Gy in 2 GY fractions on days 22 -71.
  Interventions: Drug: Irinotecan; Drug: Cisplatin

INTERVENTIONS:
Drug: Irinotecan
  Other Names: Camptosar; camptothecin-11; CPT-11
Drug: Cisplatin
  Other Names: Platinol; CDDP

SUMMARY:
This is a prospective, single institution phase II study, whose primary objective is to estimate the median and three year survival rate of non-small lung cancer patients with Stage IIIA and IIIB intra-thoracic disease which is referred to as "locally advanced" non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Patients with histological documented non-small cell lung cancer, that are considered to be inoperable, meet all the eligibility criteria, and sign informed consent will be treated with one cycle of irinotecan and cisplatin, followed by three additional cycles of chemotherapy with 60 - 70 Gy of concurrent radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documented NSCLC, including squamous cell carcinoma, adenocarcinoma, large cell carcinoma including large cell neuroendocrine carcinoma adenosquamous and sarcomatoid carcinomas.
* Patients with Pancoast tumors adjacent to a vertebral body are eligible as long as all gross disease can be encompassed in the radiation boost field. Pancoast tumor patients will be so-noted in the registry.
* Patients must be ≥ 18 years of age.
* Patients with Zubrod (ECOG) performance status ≤ 2.
* Adequate hematologic function defined as: ANC ≥ 1000/mm3, platelets ≥ 75,000/mm3, and hemoglobin ≥ 8 g/dL (prior to transfusions); adequate hepatic function defined as: total bilirubin ≤ 3.0 mg/dl, and adequate renal function defined as a serum creatinine level ≤ 2.0 mg/dl.
* Patients with weight loss ≤ 20% over the past 3 months.
* Patients with a pleural effusion that is proven cytologically negative or is too small to tap.
* Women of childbearing potential must agree to practice effective contraception throughout the study and for four weeks after completion of treatment.
* Pretreatment evaluations required for eligibility include:

  * A medical history, physical examination, and assessment of Zubrod performance status within 4 weeks prior to study entry.
  * CBC with differential and platelet count, and laboratory profile must be completed within 4 weeks prior to study entry.
  * CT scan of the chest or whole body PET (preferred), and a CT scan or MRI (preferred) of the brain within 4 weeks prior to study entry.
  * For women of childbearing potential, a serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) must be performed within a week prior to the start of protocol treatment.
  * Medical Oncology and Radiation Oncology consultation and approval.
* Patients must sign a study-specific consent form prior to study entry.

Exclusion Criteria:

* Small cell carcinomas or carcinoid histology.
* History of any malignancy in the past 2 years except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other in situ cancers.
* Prior systemic chemotherapy or radiotherapy that would interfere with delivery of treatment as outlined above as judged by the clinician.
* Cytologically malignant effusions.
* Radiographic evidence of metastatic disease.
* Active pulmonary infection not responsive to antimicrobial therapy.
* History of significant or symptomatic interstitial pneumonitis.
* Significant symptomatic cardiac disease, for example, unstable angina, uncompensated congestive heart failure, or uncontrolled cardiac ventricular arrhythmias.
* Patients with > grade 2 neuropathy.
* Women who are pregnant or breast feeding, as treatment involves unforeseeable risks to the participant, embryo, fetus, or nursing infant; women with a positive pregnancy test on enrollment or prior to study drug administration.
* Women of childbearing potential who are unwilling to practice effective contraception throughout the study and for four weeks after completion of treatment.
* Patients who currently are participating in other clinical trials and/or who have participated in other clinical trials in the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-10; Primary Completion 2017-09-27 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
Estimate the median and three year survival rate of locally advanced NSCLC using the platinum doublet cisplatin and irinotecan | Three years after the last patient has completed treatement
Estimate the progression-free survival | Three years after the last patient has completed treatement.

SECONDARY OUTCOMES:
Compare the survival of patients treated with cisplatin/irinotecan with historical controls using cisplatin/etoposide. | Three years after the last patient has completed treatment.
Measure toxicities and compliance of patients on this regimen | Thirty days after completing treatment, averaging 100 days.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Walker, MD, FACP, Principal Investigator — Brody School of Medicine at East Carolina University
Locations (1):
- Leo W Jenkins Cancer Center, Greenville, North Carolina, United States